CLINICAL TRIAL: NCT05719675
Title: Efecto de un Programa de atención Para la Salud Sobre la Adherencia al Tratamiento en Personas Con Diabetes Mellitus Tipo 2 de Reciente diagnóstico
Brief Title: Healthcare Intervention Program on Treatment Adherence in People With Newly Diagnosed Type 2 Diabetes Mellitus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, José Fernando Mora Romo, Principal Investigator, Universidad Nacional Autonoma de Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 522006894; CE/FESI/052022/1519 (Other: Ethics committee of the Iztacala School of Higher Education.); 1012331 (Other Grant/Funding Number: Consejo Nacional de Ciencia y Tecnología)
Record Dates: First submitted 2023-01-30; First posted 2023-02-09 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Treatment Adherence; Quality of Life; Glucose Metabolism Disorders (Including Diabetes Mellitus)
Keywords: Health Psychology; Behavioral Contingencial Analysis; Treatment Adherence; Glycemic Control; Health-Related Quality of Life
MeSH Terms: conditions — Treatment Adherence and Compliance; Glucose Metabolism Disorders | interventions — Methods

STUDY DESIGN:
Intervention Model Description: The intervention will focus on three phases: (1) Dispositional alteration, where the aim will be to achieve an awareness of the disease by altering any of the factors that give rise to the performance of behaviors that interfere with adherence to treatment; (2) Alteration of one's own behavior, which would be focused on the development of healthy habits consistent with the indications of the health team for the proper management of the disease; and (3) Alteration of others' behaviors, focused on the development of skills in participants so they can alter the behaviors of significant others by means of health promotion strategies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): A healthcare model for people with Type 2 Diabetes Mellitus, based on Contingency Behavioral Analysis (CBA). The CCA model was constructed in a Mexican population by Ribes et al. (1986), and later operationalized in manuals by Rodriguez (2002). It has proven to be a suitable alternative for working with people with T2DM (Ocampo et al., 2017; Rodriguez et al., 2015; Rodriguez et al., 2016; Rivera et al., 2008; Rodriguez et al., 2013; Rosales et al., 2021). For this intervention, an application manual aimed at the intervention facilitator was developed and evaluated by a panel of experts in the field of nursing, endocrinology, diabetology and social work with experience in the care of people with T2DM. In general, they were asked to evaluate the congruence and adequacy of the activities proposed in the sessions to improve adherence to treatment in people with T2DM. Additionally, they evaluated whether the number of sessions was adequate for the objectives of the research project.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — The general outline of the intervention is divided into three phases:
  1. Dispositional alteration, where the aim will be to obtain precise information on the barriers that patients encounter in carrying out their treatment and thus focus the issues to achieve an awareness of the disease by altering some of the factors that give rise to the realization of behaviors that interfere with treatment adherence.
  2. Alteration of one's own behavior, focused on the development of healthy habits that are consistent with the indications of the health team for the proper management of the disease.
  3. Alteration of the behavior of others, focused on the development of skills in the participants so that they are able to modify the behavior of other people close to them through health promotion strategies.
  Other Names: Contingency Behavioral Analysis

SUMMARY:
Type 2 Diabetes Mellitus (T2DM) is a group of metabolic disorders characterized by hyperglycemia in the absence of treatment, positioned in the first places of prevalence and mortality in the Mexican population. Adherence to treatment is a central element to prevent complications of the disease, where the active participation of the patient in his or her treatment is fundamental. Despite institutional healthcare efforts to promote this element, there is no clarity in the Clinical Practice Guidelines aimed at the attention of people with T2DM on how to achieve it.

The aim of this project will be to evaluate the effect of an intervention based on Contingency Behavior Analysis on treatment adherence, quality of life and glycemic level in people with newly diagnosed T2DM.

Pre-experimental design with pretest and posttest measurements. The Dependent Variable will be an intervention based on Contingency Behavior Analysis.

The Independent Variables will be adherence to treatment, quality of life and glycemic level.

The power calculation suggests an n = 38, using sequential non-probability sampling.

People older than 18 years with less than 5 years of T2DM diagnosis will be included.

Pretest and posttest differences, effect size and correlations between measurement variables will be analyzed.

It is expected that the intervention based on Contingency Behavior Analysis will encourage the active participation of people with T2DM, improving their adherence to treatment, glycemic level and quality of life.

Considering that the Clinical Practice Guidelines emphasize the importance of therapeutic adherence through the active participation of the patient and his/her environment, it is expected that this project will provide the tools for behavioral change that so far are not included in public health in Mexico.

DETAILED DESCRIPTION:
Currently, Type 2 Diabetes Mellitus (T2DM) in Mexico is the third leading cause of mortality in men and the second leading cause in women. Furthermore, due to the inadequate management of T2DM during the Covid-19 pandemic, an excess mortality of 35.6% was observed in the January-August 2020 period. The impact of the disease on people's health is also reflected in morbidity through diabetic complications and comorbidities related to T2DM such as cardiovascular diseases, dyslipidemias, overweight and obesity. In the case of diabetic comorbidities and complications it must be considered that sometimes they are not really due to inadequate self-care on the part of the patient, but are part of the natural progression of the disease as each person ages. However, whether the origin of diabetic complications is due to the patient's inadequate self-care behaviors or to the natural progression of the disease, the person with T2DM needs to receive comprehensive guidance to cope with disease conditions, treatment and self-care through prevention strategies and diabetes education.

In this regard, over the last decade, the Mexican health system has made various efforts to address this issue. Either through national health care programs at the federal and state levels, or through the implementation of mexican Clinical Practice Guidelines (mCPG) for the management of patients with T2DM. However, despite these implementations, in a period of 9 years (2011-2020) an increase in the registered death rate due to T2DM has been observed from 7.0 per ten thousand inhabitants in 2011 to 8.2 in 2020, which suggests that a change in the practice of care directed to this population is necessary. Perhaps one of the main problems that prevents a change in practice is the belief that it is enough to simply provide people with information on health care so that they are able to implement it in their daily lives. However, for years it has been pointed out and demonstrated that this was not enough, but that it was also necessary to provide people with the appropriate strategies for the development of new care behaviors. To achieve this, the Latin American Diabetes Association has recommended that programs encourage the active participation of people with T2DM, a recommendation that is even reflected in some health programs in Mexico . This leads to the second problem that is hindering the development of true health care that fosters the active participation of its users: professional training. In Mexico, the psychology professional is considered as a healthcare provider only on the rehabilitation of the adult lower extremity amputee patient due to T2DM, in the follow-up of physical exercise prescription, as part of nursing interventions for the control of T2DM in adult population, and in the prevention and diagnosis of T2DM in pediatric patients. This occurs despite the fact that most programs and mCPGs emphasize the importance of psychological assessment and intervention for the modification of risk behaviors and the development of healthy habits. However, by not considering psychology professionals formally to carry out education strategies, these tasks are relegated to other professionals such as physicians, nurses, nutritionists and social workers who, although they have the training to provide information about diabetes, do not have adequate training to promote the necessary behavioral modification in the development of healthy habits and promote the active participation of patients with T2DM in the search for solutions to contextual barriers, promoting health care in their daily lives through deprofessionalization work.

It would be expected that this intervention model, by improving the TA of people with Type 2 Diabetes Mellitus, would improve the participants' evaluation of their quality of life in areas such as diabetes control, anxiety related to the disease, social burden, sexual function and energy, as well as in glycemic level, mainly. In addition, this type of intervention proposals can offer a double benefit in terms of Effectiveness by modifying those situational aspects that hinder an adequate adherence to treatment in people with T2DM; and in terms of Efficiency, by allowing to carry out a work where participants can be trained as health promoters, and thus increase the dissemination of health services through the mediation of participants in the sectors close to them and that, due to institutional limitations, this population does not have direct access to them.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age.
2. Have less than 5 years with the diagnosis of Diabetes Mellitus Type 2.
3. Ability to be present for 60-90 minutes in face-to-face sessions.
4. Additionally, since it is common for people with T2DM to have several comorbidities, this study will include people who also have hypertension, overweight/obesity or dyslipidemia, since in the National Health Survey (INSP, 2021) these were considered to be the comorbidities with the greatest impact at the national level.

Exclusion Criteria:

1. Having any present complication derived from poor diabetes control such as neuropathy, retinopathy, nephropathy or lower limb amputations due to poor control of the disease. This is due to the fact that the intervention is inserted within a secondary prevention scheme, where the aim is for people with T2DM to reduce the risk of developing complications (Seguí et al., 2011).
2. Refusal by the participant to attend the intervention sessions.
3. Having a psychological or psychiatric disorder diagnosed by a health professional that prevents active participation in the workshops.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Treatment adherence | 3 months
  The Therapeutic Adherence scale for patients with chronic diseases based on explicit behaviors (Soria et al., 2009) will be used. The instrument has 21 items where the answers are presented on a scale of 0 to 100 points, considering that a person presents good adherence to treatment the closer to 100. Originally, the total scale was constructed and validated in the Mexican population, where it presented a Cronbach's Alpha of .919, and this reliability coefficient ranged between .883 and .902 for each of its items. Regarding the dimensions that make up the scale, the authors report three factors: Control over medication and food intake (α= .877), Behavioral medical follow-up (α= .798) and Self-efficacy (α= .850). The first refers to monitoring medication intake and adherence to diet; the second refers to long-term health care behaviors, such as attendance at follow-up visits; and the third factor measures the person's belief that what he does has a positive impact on his or her health.
Fasting glucose | 3 months
  An Accu-Chek Active capillary glucose kit calibrated for plasma measurements and designed to be used on the outside of the body (finger, palm or forearm) will be used.
Health-related quality of life | 3 months
  The validated version of the Diabetes-39 questionnaire (López-Carmona and Rodríguez-Moctezuma, 2006) will be used in Mexican patients. The questionnaire contains 39 items grouped into five sections: Energy and Mobility (α = .92), Diabetes Control (α = .83), Anxiety-Concern (α = .80), Social Burden (α = .83), and Sexual Functioning (α = .93). For its part, the total questionnaire had a high reliability (α = .95). Participants answer on a scale of 1 to 7 how much, in the last month, their quality of life has been affected based on the activities posed along each item, where a higher score reflects a greater affectation. In addition, it contains two final items where the patient's perception of his or her overall quality of life and the severity of diabetes is rated. The minimum values of the scale start with 0 points and reach a maximum of 100 points, where higher values indicate a greater affectation to the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Georgina E Bazán-Riverón, Study Director — Universidad Nacional Autonoma de Mexico
Locations (1):
- Facultad de Estudios Superiores Iztacala, Universidad Nacional Autónoma de México., Estado de México, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on request to the authors of the research project.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact j_fmora@hotmail.com